CLINICAL TRIAL: NCT04009642
Title: Cardiac Rest and Stress Metabolism in Patients With Type 2 Diabetes - The CardioMET Study
Brief Title: Cardiac Rest and Stress Metabolism in Patients With Type 2 Diabetes
Acronym: CardioMET
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0633
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Cardiomyopathy; Metabolic Disturbance; Fatty Acid Oxidation Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetes
  Interventions: Other: Surely observational based on disease state
- Non Diabetic
  Interventions: Other: Surely observational based on disease state

INTERVENTIONS:
Other: Surely observational based on disease state — Metabolism in T2DM vs non diabetic

SUMMARY:
The number of people with diabetes is rising. One of the major causes of premature death in diabetes is heart failure (HF). This is when the heart cannot pump blood effectively, and this may be related to abnormalities in energy production in the heart muscle. In healthy people, the heart muscle cells show flexibility and can use both sugar and fat molecules for energy production. Although burning fat provides more energy, this process requires more oxygen than burning sugars. As a result, fat is a less efficient fuel for the heart compared to sugars, especially in situations where the energy and oxygen needs are higher, such as during exercise. The investigators propose that the heart muscle in patients with type 2 diabetes relies heavily on fat for energy provision, and fails to burn more sugar molecules for energy provision during exercise to more efficiently use oxygen. Fat and sugar uptake by the heart can be detected by the difference between the blood sugar and fat levels delivered to the heart and returning from the heart, both at rest and also when the heart is working faster during Dobutamine infusion. Dobutamine is a drug frequently used to mimic exercise, and get the heart running faster during medical tests. To test the hypothesis, the investigators will assess fat and sugar uptake by the heart at rest and when the heart is running faster, in patients with type 2 diabetes undergoing investigations to rule out coronary disease. Heart function, and blood supply to heart muscle, at rest and during Dobutamine infusion, will also be measured using MRI scanning. The same tests will be performed in people without diabetes for comparison. It will help understand diabetic heart disease and which aspects may be targeted with new treatments.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Type 2 diabetes cohort:

1. Participant is willing and able to give informed consent for participation in the study.
2. Aged 18 years or above.
3. Confirmed diagnosis of T2D according to World Health Organisation (WHO) criteria
4. Undergoing invasive coronary angiography for exclusion of CAD.
5. Able (in the investigator's opinion) and willing to comply with all study requirements
6. Must understand written and verbal English

Group 2: Non-diabetic Controls

1. Participant is willing and able to give informed consent for participation in the study.
2. Aged 18 years or above.
3. Undergoing invasive coronary angiography for exclusion of CAD.
4. Able (in the investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria:

Group 1

1. Type 1 diabetes.
2. Significant CAD> (50% luminal stenosis)
3. Significant renal impairment (eGFR<30ml/min/m2).
4. Previous coronary artery bypass grafting surgery or myocardial infarction
5. Significant clinical established diagnosis of heart failure and EF <40%
6. Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
7. Participants who have participated in another research study involving an investigational product in the past 12 weeks
8. Atrial fibrillation.
9. Contra-indications to magnetic resonance imaging (pacemaker, cranial aneurysm clips, metallic ocular foreign bodies, severe claustrophobia).
10. Known hypersensitivity to dobutamine or gadolinium.
11. Participants with a diagnosis of significant (>moderate,) valve disease.

1. Patients who are on Insulin therapy, or oral Thiazolidinedione. 2. Involvement in other studies thought to compromise resulting study data or the health of the participant in the opinion of investigator.

Group 2

1. As per group 1 plus
2. Diagnosis of diabetes or impaired glucose tolerance Note patients with previous CAD treated by angioplasty/stenting and no residual disease are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1. Patients with T2D and no significant CAD (<50% luminal stenosis on coronary angiography) Group 2. Non-diabetic individuals with no significant CAD (<50% luminal stenosis on coronary angiography)
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The difference in myocardial FA extraction fraction (%) between T2D patients and non-diabetic controls at rest. | Immediate at rest and stress
  Myocardial extraction fraction

CONTACTS AND LOCATIONS:
Locations (1):
- Glenfield Hospital, University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No